CLINICAL TRIAL: NCT03899844
Title: Blood Amyloid-Beta Relationship With Amyloid Plaques and CSF Amyloid-Beta
Brief Title: Study to Evaluate Amyloid in Blood and Imaging Related to Dementia
Acronym: SEABIRD
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201902081
Record Dates: First submitted 2019-03-22; First posted 2019-04-02 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Alzheimer Disease; Alzheimer Dementia
MeSH Terms: conditions — Alzheimer Disease | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cognitively normal: 896 of the 1120 enrolled will not exhibit subjective impairment as defined by a brief clinical test. These participants will complete an initial blood collection and cognitive testing, and a subset of participants will be asked to return for a larger blood collection, amyloid (PiB) PET imaging, and MRI.
  Interventions: Other: Blood collection, PiB PET/MRI, and cognitive testing
- Cognitively impaired: 224 of the 1120 enrolled will exhibit subjective impairment as defined by a brief clinical test. These participants will complete an initial blood collection and cognitive testing, and a subset of participants will be asked to return for a larger blood collection, amyloid (PiB) PET imaging, and MRI.
  Interventions: Other: Blood collection, PiB PET/MRI, and cognitive testing

INTERVENTIONS:
Other: Blood collection, PiB PET/MRI, and cognitive testing — Blood and imaging results will be analyzed for amyloid beta. Cognitive testing will be performed to determine clinical and cognitive status.

SUMMARY:
The purpose of this study is to determine how well a blood test can detect amyloid beta, a protein involved in Alzheimer's disease. Participants will be asked to complete an initial blood collection and cognitive testing, and a subset of participants will be asked to complete a larger blood collection, amyloid PET imaging, and an MRI.

DETAILED DESCRIPTION:
Alzheimer's disease is the most common cause of dementia and currently has no disease-modifying treatments or simple, accurate diagnostic tests. Amyloid beta builds up in the brain and forms plaques in people with Alzheimer's disease, and the buildup of this protein is found decades before symptoms of dementia begin. A blood test may be able to quickly and inexpensively screen people for Alzheimer's disease clinical trials and eventually diagnose Alzheimer's disease in the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. At least 60 years of age

Exclusion Criteria:

1. Unable to perform one or more activities of daily living (eating, bathing, dressing, ambulating, toileting) due to cognitive impairment or dependent on others due to cognitive impairment.
2. Body weight of <100 pounds
3. Active infectious disease (e.g., HIV, hepatitis B, hepatitis C)
4. Bleeding disorder
5. Taking an experimental drug for AD
6. Blood donation in the last two months
7. Blood transfusion in the last three months
8. On hospice

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from clinics and communities throughout the greater St. Louis metropolitan area.
Sampling Method: Non-Probability Sample
Enrollment: 1122 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Plasma amyloid-beta 42/40 ratio | Baseline
Plasma amyloid-beta 42/40 ratio | 6 months
Area under the curve (AUC) of the blood test (plasma amyloid-beta 42/40 ratio) in predicting amyloid PET status | 6 months

SECONDARY OUTCOMES:
Coefficient of variation for the initial and confirmatory blood amyloid-beta test results | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Randall Bateman, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data which documents, supports and validates research findings will be made available after the main findings from the final research data set have been accepted for publication. Such research data will be de-identified to prevent the disclosure of personal identifiers.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available immediately following publication with no end date.
Access Criteria: Qualified researchers who provide a methodologically sound proposal will be able to access the data to achieve aims in the approved proposal. Proposals should be directed to batemanr@wustl.edu. To gain access, requestors will need to sign a data access agreement.